CLINICAL TRIAL: NCT01401582
Title: Dementia: Life- and Personcentered Help in Germany
Brief Title: Intervention Study to Improve Life and Care for People With Dementia and Their Caregivers in Primary Care
Acronym: DelpHi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Collaborators: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, René Thyrian, Research Group Leader, German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DZNE_DelpHi-MV_001
Record Dates: First submitted 2011-07-18; First posted 2011-07-25 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: health care; dementia care; caregiver support; epidemiological study
MeSH Terms: conditions — Dementia | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- care as usual (No Intervention): care as usual, no intervention, just observation of natural change/ trajectories over time
- Implementation of Dementia Care Manager (Experimental): Subjects in this arm will be provided with a specialised "Dementia Care Manager" to be included in a subsidiary support system
  Interventions: Other: Implementation of Dementia Care Manager

INTERVENTIONS:
Other: Implementation of Dementia Care Manager — Home-visits of trained "Dementia Care Manager (DCM)" at least monthly for 6 months. The DCM will, in close cooperation with the general practitioner, establish and include a subsidiary support system for subjects and their caregivers.
  Other Names: Dementia Care Manager; Care Management; counselling; supporting caregivers
  Arms: Implementation of Dementia Care Manager

SUMMARY:
Caring for people with dementia and treating them is a major challenge for the health care system in Germany. Among the challenges for population-based health care research are (a) identification and early recognition, (b) multimorbidity and (c) the integration of persons with dementia into the health care system. One setting which is identified to meet the challenges is the primary care setting and there especially the general physician. There have been a few interventional studies, which have been restricted to selective samples and have been conducted in inpatient settings.

The purpose of this study is to test the efficacy of implementing a subsidiary support system for persons with dementia living at home. This subsidiary support system is initiated by a Dementia Care Manager (DCM), a nurse with dementia-specific advanced training. The main goals are to improve quality of life and health care of the person with dementia and reduce caregiver´s burden.

The study is a general physician based cluster-randomised controlled intervention trial. A population based sample of general physicians will be asked to participate in a systematic screening trial to identify people with dementia in primary care in Mecklenburg Western Pommerania (MV), a federal state in Germany. Upon identification the people will be asked to participate in the DelpHi-MV study and after having given written informed consent will then be assigned to an intervention and a control group. Identification of people with dementia will be achieved by a short screening questionnaire in the physician's office. An extended in-depth data assessment will be conducted after inclusion into the study and then annually to measure the course of the people's health. Data assessment will be done at the people's homes.

People assigned to the intervention group will receive an intervention provided by "Dementia Care Manager". The Dementia Care Manager is a specialised nurse that is going into the person's home to manage the care of dementia as well as caring for the person's relative/ or carer.

DETAILED DESCRIPTION:
The "Dementia: life- and person-centered help in Mecklenburg-Western Pomerania (DelpHi)" trial was a pragmatic, general practitioner (GP)-based, cluster-randomized intervention study with two arms, an intervention group and a care as usual (CAU) group. T The design, eligibility and inclusion criteria, intervention and baseline characteristics of the trial have been described in detail elsewhere.

To reduce the risk of contamination across groups, GP practices were the unit of randomization and determined the patients´ group status. At the beginning of the study, a total of 854 GPs in 5 municipalities of Mecklenburg-Western Pomerania were invited to participate by mail. GPs expressing an interest in the study were visited by the investigators to convey additional detailed information about the study. Finally, 136 GPs (16%) gave written informed consent (IC) to participate and agreed to adhere to the DelpHi-study protocol. There were no restrictions regarding the GPs' treatment of patients.

GPs systematically assessed the eligibility of patients for the trial during routine care (eligibility criteria for screening: age >70 years, living at home). Patients were screened using screening procedure. This individual interview-based instrument is widely used for dementia screening in GP practices in Germany. Patients who screened positive were informed about the study by their GP, invited to participate and asked to provide written IC. If the patients listed a caregiver, he or she was asked to participate as well. When patients were unable to provide written IC, their legal representative was asked to sign the consent form on their behalf. The study physicians received allowances for performing the screening (10€ per patient) and study enrollment (100€ per patient).

Identical, standardized, computer-assisted face-to-face interviews with all participants were conducted at the participants' homes by specifically trained nurses over an average of three separate visits (1) immediately after study inclusion (baseline) and (2) 12 months later (follow-up). To minimize participant burden, the assessment sessions were restricted to one hour.

Dementia Care Management is a complex intervention that aims to provide "optimal care" by integrating multi-professional and multimodal strategies for improving patient- and caregiver-related outcomes. DCM individualizes and optimizes dementia treatment and care within the framework of the established health care and social service system. It was developed according to current guidelines targeted at the individual participant level and delivered at participants´ homes by 6 nurses with dementia-specific training. Nurses were supported by a computer-based intervention-management system (IMS) to improve systematic identification of patients' and caregivers' unmet needs and the subsequent recommendation of interventions to address these needs. The training as well as software are described in more detail elsewhere.

The primary outcomes pertain to the individual participants: (a) Quality of life, measured by the Quality of Life in Alzheimer's Disease instrument (QolAD); (b) Caregiver burden, measured by the "Berlin Inventory of Caregivers' Burden with Dementia Patients (BIZA-D)"; (c) Behavioral and psychological symptoms, measured by the Neuropsychiatric Inventory (NPI); (d) Use of pharmacotherapy with antidementia drugs, which included the following substances recommended by relevant guidelines: donepezil, galantamine, rivastigmine, and memantine; and (e) Use of potentially inadequate medication (PIM), evaluated using the Priscus criteria..

Sample size: No previous data on the main outcome measures were available to use for sample size calculation. Therefore, sample size was estimated based on theoretical assumptions. In the design, the minimally important difference (MID) for determining the efficacy was considered to be of at least a small effect, defined by Cohen's d (d = 0.2 48). Comparing two groups at a significance level of α = 0.05, assuming a statistical power of 80% and an intra-class correlation with clustering by GP practice of zero a sample size of 310 persons per group would have been sufficient 48. Considering the longitudinal design, we accounted for a loss over time of 35% (death, withdrawal of IC) and determined that 477 persons per group with complete datasets would have been needed to be included in the study. We estimated that GPs would identify n=1,000 participants over the course of 2 years. Recruitment turned out to be slower than expected. Thus recruitment was prolonged from two to three years. The sample size achieved allows to detect a medium effect size (Cohen´s d=0.5) 48.

Randomization/allocation We used simple 1:1 randomization without stratification or matching. This procedure was sufficient due to the high number of expected clusters in our study 49. GPs were not informed of their randomization status. However, due to the type of intervention, GPs became aware of their status throughout the course of the study. Participants were recruited and enrolled by participating GPs but allocated to the study group by study center. Since baseline assessment and delivery of intervention needed to be performed by the same nurses, a blinding was not possible.

ELIGIBILITY:
Inclusion Criteria:

* 70+ years
* must be living at home
* screening positive (DEMTECT < 9), indicating dementia

Exclusion Criteria:

* medical conditions not allowing testing

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 634 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hoffmann, MD, MPH, Principal Investigator — University Medicine Greifswald
Locations (1):
- Institute for Community Medicine, Greifswald, Mecklenburg- Western Pommerania, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Cummings JL. The Neuropsychiatric Inventory: assessing psychopathology in dementia patients. Neurology. 1997 May;48(5 Suppl 6):S10-6. doi: 10.1212/wnl.48.5_suppl_6.10s. PMID 9153155
- [Background] Erzigkeit H, Lehfeld H, Pena-Casanova J, Bieber F, Yekrangi-Hartmann C, Rupp M, Rappard F, Arnold K, Hindmarch I. The Bayer-Activities of Daily Living Scale (B-ADL): results from a validation study in three European countries. Dement Geriatr Cogn Disord. 2001 Sep-Oct;12(5):348-58. doi: 10.1159/000051280. PMID 11455136
- [Background] Fiss T, Ritter CA, Alte D, van den Berg N, Hoffmann W. Detection of drug related problems in an interdisciplinary health care model for rural areas in Germany. Pharm World Sci. 2010 Oct;32(5):566-74. doi: 10.1007/s11096-010-9409-6. Epub 2010 Jul 1. PMID 20593238
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Sandholzer H, Hellenbrand W, Renteln-Kruse W, Van Weel C, Walker P. [STEP--standardized assessment of elderly people in primary care]. Dtsch Med Wochenschr. 2004 Dec 10;129 Suppl 4:S183-226. doi: 10.1055/s-2004-836107. German. PMID 15592957
- [Background] Wimo A, Nordberg G, Jansson W, Grafstrom M. Assessment of informal services to demented people with the RUD instrument. Int J Geriatr Psychiatry. 2000 Oct;15(10):969-71. doi: 10.1002/1099-1166(200010)15:103.0.co;2-9. No abstract available. PMID 11044880
- [Background] Bullinger M, Kirchberger I. SF-36 Fragenbogen zum Gesundheitszustand. Göttingen 1998: Hogrefe-Verlag GmBH & Co.KG; 1998
- [Background] Fydrich T, Sommer G, Brähler E. F-SozU. Fragebogen zur sozialen Unterstützung. Göttingen: Hogrefe; 2007.
- [Background] Zank S, Schacke C, Leipold B. Berliner Inventar zur Angehörigenbelastung - Demenz (BIZA-D). Zeitschrift für Klinische Psychologie und Psychotherapie 2006; 35(4):296-305.
- [Background] Monsch AU. [Neuropsychological examination in evaluating dementia]. Praxis (Bern 1994). 1997 Aug 27;86(35):1340-2. German. PMID 9381025
- [Result] Reiner K, Eichler T, Hertel J, Hoffmann W, Thyrian JR. The Clock Drawing Test: A Reasonable Instrument to Assess Probable Dementia in Primary Care? Curr Alzheimer Res. 2018;15(1):38-43. doi: 10.2174/1567205014666170908101822. PMID 28891446
- [Result] Eichler T, Thyrian JR, Hertel J, Richter S, Michalowsky B, Wucherer D, Dreier A, Kilimann I, Teipel S, Hoffmann W. Patient Variables Associated with the Assignment of a Formal Dementia Diagnosis to Positively Screened Primary Care Patients. Curr Alzheimer Res. 2018;15(1):44-50. doi: 10.2174/1567205014666170908095707. PMID 28891445
- [Result] Wucherer D, Thyrian JR, Eichler T, Hertel J, Kilimann I, Richter S, Michalowsky B, Zwingmann I, Dreier-Wolfgramm A, Ritter CA, Teipel S, Hoffmann W. Drug-related problems in community-dwelling primary care patients screened positive for dementia. Int Psychogeriatr. 2017 Nov;29(11):1857-1868. doi: 10.1017/S1041610217001442. Epub 2017 Aug 7. PMID 28780910
- [Result] Thyrian JR, Hertel J, Wucherer D, Eichler T, Michalowsky B, Dreier-Wolfgramm A, Zwingmann I, Kilimann I, Teipel S, Hoffmann W. Effectiveness and Safety of Dementia Care Management in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Oct 1;74(10):996-1004. doi: 10.1001/jamapsychiatry.2017.2124. PMID 28746708
- [Result] Dreier-Wolfgramm A, Michalowsky B, Austrom MG, van der Marck MA, Iliffe S, Alder C, Vollmar HC, Thyrian JR, Wucherer D, Zwingmann I, Hoffmann W. Dementia care management in primary care : Current collaborative care models and the case for interprofessional education. Z Gerontol Geriatr. 2017 May;50(Suppl 2):68-77. doi: 10.1007/s00391-017-1220-8. Epub 2017 Mar 31. PMID 28364258
- [Result] Michalowsky B, Flessa S, Eichler T, Hertel J, Dreier A, Zwingmann I, Wucherer D, Rau H, Thyrian JR, Hoffmann W. Healthcare utilization and costs in primary care patients with dementia: baseline results of the DelpHi-trial. Eur J Health Econ. 2018 Jan;19(1):87-102. doi: 10.1007/s10198-017-0869-7. Epub 2017 Feb 3. PMID 28160100
- [Result] Wucherer D, Eichler T, Hertel J, Kilimann I, Richter S, Michalowsky B, Thyrian JR, Teipel S, Hoffmann W. Potentially Inappropriate Medication in Community-Dwelling Primary Care Patients who were Screened Positive for Dementia. J Alzheimers Dis. 2017;55(2):691-701. doi: 10.3233/JAD-160581. PMID 27716668
- [Result] Thyrian JR, Winter P, Eichler T, Reimann M, Wucherer D, Dreier A, Michalowsky B, Zarm K, Hoffmann W. Relatives' burden of caring for people screened positive for dementia in primary care : Results of the DelpHi study. Z Gerontol Geriatr. 2017 Jan;50(1):4-13. doi: 10.1007/s00391-016-1119-9. Epub 2016 Aug 17. PMID 27534949
- [Result] Eichler T, Thyrian JR, Hertel J, Wucherer D, Michalowsky B, Reiner K, Dreier A, Kilimann I, Teipel S, Hoffmann W. Subjective memory impairment: No suitable criteria for case-finding of dementia in primary care. Alzheimers Dement (Amst). 2015 Apr 30;1(2):179-86. doi: 10.1016/j.dadm.2015.02.004. eCollection 2015 Jun. PMID 27239503
- [Result] Thyrian JR, Eichler T, Pooch A, Albuerne K, Dreier A, Michalowsky B, Wucherer D, Hoffmann W. Systematic, early identification of dementia and dementia care management are highly appreciated by general physicians in primary care - results within a cluster-randomized-controlled trial (DelpHi). J Multidiscip Healthc. 2016 Apr 19;9:183-90. doi: 10.2147/JMDH.S96055. eCollection 2016. PMID 27143912
- [Result] Thyrian JR, Eichler T, Michalowsky B, Wucherer D, Reimann M, Hertel J, Richter S, Dreier A, Hoffmann W. Community-Dwelling People Screened Positive for Dementia in Primary Care: A Comprehensive, Multivariate Descriptive Analysis Using Data from the DelpHi-Study. J Alzheimers Dis. 2016 Mar 30;52(2):609-17. doi: 10.3233/JAD-151076. PMID 27031481
- [Result] Eichler T, Hoffmann W, Hertel J, Richter S, Wucherer D, Michalowsky B, Dreier A, Thyrian JR. Living Alone with Dementia: Prevalence, Correlates and the Utilization of Health and Nursing Care Services. J Alzheimers Dis. 2016;52(2):619-29. doi: 10.3233/JAD-151058. PMID 27031480
- [Result] Eichler T, Thyrian JR, Hertel J, Richter S, Wucherer D, Michalowsky B, Teipel S, Kilimann I, Dreier A, Hoffmann W. Unmet Needs of Community-Dwelling Primary Care Patients with Dementia in Germany: Prevalence and Correlates. J Alzheimers Dis. 2016;51(3):847-55. doi: 10.3233/JAD-150935. PMID 26890767
- [Result] Thyrian JR, Eichler T, Reimann M, Wucherer D, Dreier A, Michalowsky B, Hoffmann W. Depressive symptoms and depression in people screened positive for dementia in primary care - results of the DelpHi-study. Int Psychogeriatr. 2016 Jun;28(6):929-37. doi: 10.1017/S1041610215002458. Epub 2016 Jan 20. PMID 26785854
- [Result] Michalowsky B, Thyrian JR, Eichler T, Hertel J, Wucherer D, Flessa S, Hoffmann W. Economic Analysis of Formal Care, Informal Care, and Productivity Losses in Primary Care Patients who Screened Positive for Dementia in Germany. J Alzheimers Dis. 2016;50(1):47-59. doi: 10.3233/JAD-150600. PMID 26639964
- [Result] Michalowsky B, Eichler T, Thyrian JR, Hertel J, Wucherer D, Hoffmann W, Flessa S. Healthcare resource utilization and cost in dementia: are there differences between patients screened positive for dementia with and those without a formal diagnosis of dementia in primary care in Germany? - ERRATUM. Int Psychogeriatr. 2016 Mar;28(3):371. doi: 10.1017/S1041610215001908. Epub 2015 Oct 29. PMID 26510524
- [Result] Dreier A, Thyrian JR, Eichler T, Hoffmann W. Qualifications for nurses for the care of patients with dementia and support to their caregivers: A pilot evaluation of the dementia care management curriculum. Nurse Educ Today. 2016 Jan;36:310-7. doi: 10.1016/j.nedt.2015.07.024. Epub 2015 Jul 31. PMID 26277428
- [Result] Thyrian JR, Eichler T, Hertel J, Wucherer D, Dreier A, Michalowsky B, Killimann I, Teipel S, Hoffmann W. Burden of Behavioral and Psychiatric Symptoms in People Screened Positive for Dementia in Primary Care: Results of the DelpHi-Study. J Alzheimers Dis. 2015;46(2):451-9. doi: 10.3233/JAD-143114. PMID 25765916
- [Result] Eichler T, Thyrian JR, Hertel J, Michalowsky B, Wucherer D, Dreier A, Kilimann I, Teipel S, Hoffmann W. Rates of formal diagnosis of dementia in primary care: The effect of screening. Alzheimers Dement (Amst). 2015 Mar 29;1(1):87-93. doi: 10.1016/j.dadm.2014.11.007. eCollection 2015 Mar. PMID 27239495
- [Result] Wucherer D, Eichler T, Kilimann I, Hertel J, Michalowsky B, Thyrian JR, Teipel S, Hoffmann W. Antidementia drug treatment in people screened positive for dementia in primary care. J Alzheimers Dis. 2015;44(3):1015-21. doi: 10.3233/JAD-142064. PMID 25391382
- [Result] Teipel SJ, Thyrian JR, Hertel J, Eichler T, Wucherer D, Michalowsky B, Kilimann I, Hoffmann W. Neuropsychiatric symptoms in people screened positive for dementia in primary care. Int Psychogeriatr. 2015 Jan;27(1):39-48. doi: 10.1017/S1041610214001987. Epub 2014 Sep 23. PMID 25247664
- [Result] Eichler T, Wucherer D, Thyrian JR, Kilimann I, Hertel J, Michalowsky B, Teipel S, Hoffmann W. Antipsychotic drug treatment in ambulatory dementia care: prevalence and correlates. J Alzheimers Dis. 2015;43(4):1303-11. doi: 10.3233/JAD-141554. PMID 25147117
- [Result] Michalowsky B, Eichler T, Thyrian JR, Hertel J, Wucherer D, Laufs S, Flessa S, Hoffmann W. Medication cost of persons with dementia in primary care in Germany. J Alzheimers Dis. 2014;42(3):949-58. doi: 10.3233/JAD-140804. PMID 25125471
- [Result] Eichler T, Thyrian JR, Hertel J, Kohler L, Wucherer D, Dreier A, Michalowsky B, Teipel S, Hoffmann W. Rates of formal diagnosis in people screened positive for dementia in primary care: results of the DelpHi-Trial. J Alzheimers Dis. 2014;42(2):451-8. doi: 10.3233/JAD-140354. PMID 24898640
- [Result] Eichler T, Thyrian JR, Fredrich D, Kohler L, Wucherer D, Michalowsky B, Dreier A, Hoffmann W. The benefits of implementing a computerized intervention-management-system (IMS) on delivering integrated dementia care in the primary care setting. Int Psychogeriatr. 2014 Aug;26(8):1377-85. doi: 10.1017/S1041610214000830. Epub 2014 May 9. PMID 24811145
- [Result] Fiss T, Thyrian JR, Wucherer D, Assmann G, Kilimann I, Teipel SJ, Hoffmann W. Medication management for people with dementia in primary care: description of implementation in the DelpHi study. BMC Geriatr. 2013 Nov 13;13:121. doi: 10.1186/1471-2318-13-121. PMID 24225205
- [Result] Eichler T, Thyrian JR, Dreier A, Wucherer D, Kohler L, Fiss T, Bowing G, Michalowsky B, Hoffmann W. Dementia care management: going new ways in ambulant dementia care within a GP-based randomized controlled intervention trial. Int Psychogeriatr. 2014 Feb;26(2):247-56. doi: 10.1017/S1041610213001786. Epub 2013 Oct 23. PMID 24152974
- [Result] Thyrian JR, Fiss T, Dreier A, Bowing G, Angelow A, Lueke S, Teipel S, Flessa S, Grabe HJ, Freyberger HJ, Hoffmann W. Life- and person-centred help in Mecklenburg-Western Pomerania, Germany (DelpHi): study protocol for a randomised controlled trial. Trials. 2012 May 10;13:56. doi: 10.1186/1745-6215-13-56. PMID 22575023
- [Derived] Michalowsky B, Blotenberg I, Platen M, Teipel S, Kilimann I, Portacolone E, Bohlken J, Radke A, Buchholz M, Scharf A, Muehlichen F, Xie F, Thyrian JR, Hoffmann W. Clinical Outcomes and Cost-Effectiveness of Collaborative Dementia Care: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2419282. doi: 10.1001/jamanetworkopen.2024.19282. PMID 38967926
- [Derived] Muhlichen F, Michalowsky B, Radke A, Platen M, Mohr W, Thyrian JR, Hoffmann W. Tasks and Activities of an Effective Collaborative Dementia Care Management Program in German Primary Care. J Alzheimers Dis. 2022;87(4):1615-1625. doi: 10.3233/JAD-215656. PMID 35491783
- [Derived] Muller B, Kropp P, Cardona MI, Michalowsky B, van den Berg N, Teipel S, Hoffmann W, Thyrian JR. Types of leisure time physical activities (LTPA) of community-dwelling persons who have been screened positive for dementia. BMC Geriatr. 2021 Apr 23;21(1):270. doi: 10.1186/s12877-021-02201-1. PMID 33892624
- [Derived] Zwingmann I, Dreier-Wolfgramm A, Esser A, Wucherer D, Thyrian JR, Eichler T, Kaczynski A, Monsees J, Keller A, Hertel J, Kilimann I, Teipel S, Michalowsky B, Hoffmann W. Why do family dementia caregivers reject caregiver support services? Analyzing types of rejection and associated health-impairments in a cluster-randomized controlled intervention trial. BMC Health Serv Res. 2020 Feb 14;20(1):121. doi: 10.1186/s12913-020-4970-8. PMID 32059724
- [Derived] Zwingmann I, Michalowsky B, Esser A, Kaczynski A, Monsees J, Keller A, Hertel J, Wucherer D, Thyrian JR, Eichler T, Kilimann I, Teipel S, Dreier Wolfgramm A, Hoffmann W. Identifying Unmet Needs of Family Dementia Caregivers: Results of the Baseline Assessment of a Cluster-Randomized Controlled Intervention Trial. J Alzheimers Dis. 2019;67(2):527-539. doi: 10.3233/JAD-180244. PMID 30584136
- [Derived] Brueggen K, Dyrba M, Kilimann I, Henf J, Hoffmann W, Thyrian JR, Teipel S. Hippocampal Mean Diffusivity for the Diagnosis of Dementia and Mild Cognitive Impairment in Primary Care. Curr Alzheimer Res. 2018;15(11):1005-1012. doi: 10.2174/1567205015666180613114829. PMID 29895247
- [Derived] Zwingmann I, Hoffmann W, Michalowsky B, Wucherer D, Eichler T, Teipel S, Dreier-Wolfgramm A, Kilimann I, Thyrian JR. [Unmet needs of family dementia caregivers of persons with dementia : Primary medical care]. Nervenarzt. 2018 May;89(5):495-499. doi: 10.1007/s00115-018-0509-1. German. PMID 29619534
- [Derived] Teipel SJ, Keller F, Thyrian JR, Strohmaier U, Altiner A, Hoffmann W, Kilimann I. Hippocampus and Basal Forebrain Volumetry for Dementia and Mild Cognitive Impairment Diagnosis: Could It Be Useful in Primary Care? J Alzheimers Dis. 2017;55(4):1379-1394. doi: 10.3233/JAD-160778. PMID 27834778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1/1/2012-12/31/2014 Screening in participating General practices (GP)
Groups:
- Implementation of Dementia Care Manager: Subjects in this arm will be provided with a specialised "Dementia Care Manager" to be included in a subsidiary support system
  Provision of a "Dementia Care Manager": Home-visits of trained "Dementia Care Manager (DCM)" at least monthly for 6 months. The DCM will, in close cooperation with the general practitioner, establish and include a subsidiary support system for subjects and their caregivers.
Period: Overall Study
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Started | 226 | 408
Baseline Completed | 168 | 348
Completed | 116 | 291
Not Completed | 110 | 117

BASELINE CHARACTERISTICS:
Population: published in Thyrian et al. (2016). Journal of Alzheimer´s Disease (52); 69-617.
Groups:
- Care as Usual: care as usual, no intervention, just observation of natural change/ trajectories over time
  published in Thyrian et al. (2016). Journal of Alzheimer´s Disease (52); 69-617.
- Implementation of Dementia Care Manager: Subjects in this arm will be provided with a specialised "Dementia Care Manager" to be included in a subsidiary support system
  Provision of a "Dementia Care Manager": Home-visits of trained "Dementia Care Manager (DCM)" at least monthly for 6 months. The DCM will, in close cooperation with the general practitioner, establish and include a subsidiary support system for subjects and their caregivers.
  published in Thyrian et al. (2016). Journal of Alzheimer´s Disease (52); 69-617.
- Total: Total of all reporting groups
Arm/Group | Care as Usual | Implementation of Dementia Care Manager | Total
Number analyzed (Participants) | 168 | 348 | 516
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (5.3) | 80.2 (5.7) | 80.0 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 211 | 307
  Male | 72 | 137 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 168 | 348 | 516
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: The Quality of Life in Alzheimer's Disease (Qol-AD; Logsdon et al. 2002) was used. This measure designed specifically to obtain a rating of the patient's quality of life from both the patient and the caregiver. Each item is rated on a four point scale, with 1 being poor and 4 being excellent. Total scores, obtained by the sum of all 13 items, range from 13 to 52.
Time Frame: one year after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
units on a scale | 2.8 (0.3) | 2.8 (0.4)

2. Primary Outcome: Change in Caregiver Burden
Description: Caregiver burden was assessed using the "Berliner Inventar zur Angehörigenbelastung - Demenz" (BIZA-D) (Zank et al., 2006). The BIZAD was developed to assess objective as well as subjective burden due to caring for a person wit dementia (PWD). It consists of 88 items covering 20 dimensions of caregiver burden. Objective burden is divided into six dimensions: 1) basic care tasks like support eating, hygiene etc (7 items), 2) extended care tasks like supporting grocery shopping, legal affairs etc. (3 items), 3) Motivation and Guidance (4 items), 4) emotional support (4 items), 5) supporting maintenance of social contacts (3 items) and 6) supervision (4 items). Each item has to be rated regarding the frequency of the support needed on a 5-Point scale (example: supervision; Does the patient need this kind of support: 1=always, 2= mostly, 3=partly, 4=hardly, 5= not at all). Then each item asks: Who is providing this support: all by someone else, mostly by someone else, evenly distributed
Time Frame: one year after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
units on a scale | 0.4 (2.62) | 0.13 (2.63)

3. Primary Outcome: Change in Behavioral and Psychological Symptoms of Dementia
Description: Neuropsychiatric Inventory (NPI; Cummings 1997); The NPI represents an interview by proxy on twelve dimensions of neuropsychiatric behaviors, i.e. delusions, hallucinations, agitation, dysphoria, anxiety, apathy, irritability, euphoria, disinhibition, aberrant motor behavior, night-time behavior disturbances, and appetite and eating abnormalities. The presence (0= no, 1= yes) is asked. If present, the severity (rated 1 through 3; mild to severe) and frequency (1 to 4, rarely to very often) of each neuropsychiatric symptom are rated on. Thus the score for each dimension ranges from 0 = not present, 1= mildly and rarely to 12 = severe and often. A total NPI score is calculated as the sum of the frequency by severity scores ofeach domain range: 0 to 144, the higher the more neuropsychiatric symptomatic).
Time Frame: one year after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
units on a scale | 15.2 (16.9) | 8.2 (13.6)

4. Primary Outcome: Change in Medical Treatment With Antidementia Drugs
Description: medication was systematically reviewed; A computer-based home medication review (HMR) encompasses all medications used by the study participants and includes questions about compliance, adverse effects and drug administration. The collection of primary data on medication in the context of the HMR includes both prescription drugs and over-the-counter drugs. The assignment was then integrated using a master file of the Pharmaceutical Index. The following antidementia drugs were considered: donepezil (N06AD02), rivastigmine (N06AD03), galantamine (N06AD04) and memantine (N06AX01).
Time Frame: one year after baseline assessment
Measure: Number; unit: participants
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
participants | 31 | 114

5. Primary Outcome: Reduction of Potential Inapropriate Medication (PIM)
Description: Having to deal with multimorbidity and polypharmacy in a sample of chronically ill elderly, we also analyze potentially inappropriate medication (PIM), defined as "a drug for which the risk of an adverse event outweighs the clinical benefit, particularly when there is evidence in favor of a safer or more effective alternative therapy for the same condition". The PIM were identified using the Priscus list, which contains 83 drugs from 18 different drug classes.
Time Frame: one year after baseline assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
Participants | 19 | 77

6. Secondary Outcome: Person With Dementia: Change in Activities of Daily Living
Description: The functional status was assessed using the Bayer Activities of Daily Living Scale (B-ADL). It coonsits of 25 Items indicating everyday problems/ challenges. Their occurence is rated on a scale of 1 "never", to 10 "always". All ratings are added and divided by the number of items. This yields a mean score of 1 to 10, where 1 indicates the lowest possible impairment and 10 indicates the highest possible impairment.
Time Frame: one year after baseline assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
Number analyzed (Participants) | 116 | 291
units on a scale | 4.4 (2.4) | 4.9 (2.9)

7. Secondary Outcome: Person With Dementia: Change in Social Support
Description: The F-SozU (Fydrich et al. 2007) will be used to assess social support in several domains
Time Frame: participants will be followed yearly until institutionalisation or death after an expected average of 5 years
Reporting Status: Not Posted, anticipated posting 2026-05

8. Secondary Outcome: Person With Dementia and Caregiver: Change in Health Status
Description: Several instruments will be used to assess the health of the person with dementia:
  the GP records the Fragebogen zum SF12- health survey (SF-12, Bullinger et al. 1998) the standardized assessment of elderly in primary care (STEP; Sandholzer et al. 2004) the Brief Symptom Inventory (BSI; Derogatis et al. 1983) the Patient´s health questionnaire (PHQ-D; Löwe et al. 2002, Spitzer et al. 1999)
Time Frame: participants will be followed yearly until institutionalisation or death after an expected average of 5 years
Reporting Status: Not Posted, anticipated posting 2026-05

9. Secondary Outcome: Person With Dementia: Change in Utilization of Health Care Resources
Description: frequency of utilisation of
  1. general physicians and physicians of other specialties
  2. out-patient treatments
  3. in-patient treatments
  4. hospitalisations
  5. institutionalisation
  6. therapeutic appliances
  standardised assessment with the Resource Utilization in Dementia (RUD, Wimo et al. 1998).
Time Frame: participants will be followed yearly until institutionalisation or death after an expected average of 5 years
Reporting Status: Not Posted, anticipated posting 2026-05

10. Secondary Outcome: Person With Dementia: Change in Medication
Description: The DCM will conduct an IT-supported home medication review (Fiss et al., 2010) at the patients home with subsequent medication management by the local pharmacy regarding frequency of drug related problems, intake of PIM, clinically relevant drug-drug interaction, adherence, utilisation of adherence supporting activities (medication plan, drug dispenser, support by care service, reduction of the number of drugs taken
Time Frame: participants will be followed yearly until institutionalisation or death after an expected average of 5 years
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: over a time period of 24 months following baseline assessment
Arm/Group | Care as Usual | Implementation of Dementia Care Manager
All-Cause Mortality (participants affected / at risk) | 19/226 | 35/408
Serious Adverse Events (participants affected / at risk) | 0/226 | 0/408
Other Adverse Events (participants affected / at risk) | 0/226 | 0/408

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2016-11-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT01401582/SAP_000.pdf